CLINICAL TRIAL: NCT01692613
Title: Confocal Endomicrosopy for the Detection of Food Intolerance in Patients With Irritable Bowel Syndrome
Brief Title: Endomicroscopy, IBS and Food Intolerance
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Mark Ellrichmann, Dr., University Hospital Schleswig-Holstein
Other Study IDs: A139/12
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Endomicroscopy; Inflammatory Bowel Syndrome; Food Intolerance
MeSH Terms: conditions — Food Intolerance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * duodenal biopsies
  * duodenal fluid
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background:

The immediate endoscopic identification and diagnosis of intraepithelial structures and immediate and delayed reactions to allergens in the mucosal surface of the gut are unmet goals in the diagnosis and management of subjects with food intolerances, who are negative to all available tests. Endomicroscopy may be helpful to further visualize and characterize unmasked small bowel reactions to foods, which has not been described before.

Confocal laser endomicroscopy provides confocal microscopic imaging simultaneously to the macroscopic view ,which enables the examiner to see immediate reactions after exposure and it further allows capturing of fluid excreted by the gut for further analysis to understand the pathology behind this reaction further.

N=50 patients with unexplained bloating and diarrhoea with suspicion of food intolerance and negative testing with routine methods. Patients with Lactose intolerance n=10 patients to compare results. Patients with Fructose intolerance n=10 patients to compare results. Volunteers with Barrett's esophagus who need evaluation for possible dysplasia in the Barrett's mucosa with confocal endomicrosopy but no symptoms of bloating and abdominal pain (n=10) to serve as healthy controls for allergy testing.

Methods:

The primary objective is to investigate whether endomicroscopy will allow the detection of an allergic reaction of the gut after exposure of the 5 major allergens in the following way:

After standard gastroscopy with the endomicroscope including evaluation of the surface of the upper gastrointestinal tract, i.v. injection of Fluorescein, then initial visualisation of the duodenal surface including count of initial lymphocytes/mononuclear cells in the lamina propria: Allergen 1 (milk), allergen 2 (wheat), allergen 3 (soya),allergen 4 (apple), allergen 5 (yeast).

The primary endpoint is the visible marked increase of lymphocytes and mononuclear cells in the lamina propria of the duodenum, representing an acute reaction to one of the allergens sprayed to its surface through the endoscope channel.

DETAILED DESCRIPTION:
The primary endpoint is the visible marked increase of lymphocytes and mononuclear cells in the lamina propria of the duodenum, representing an acute reaction to one of the allergens sprayed to its surface through the endoscope channel.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* ongoing abdominal symptoms such as bloating and abdominal pain
* negative routine testing for food intolerance (or known lactose/fructose intolerance)
* written informed consent

Exclusion Criteria:

* no consent
* known reason for the abdominal pain and bloating other than lactose/fructose intolerance
* M. Whipple
* known infectious gastrointestinal disease
* stricture in the upper gastrointestinal tract
* age >18years
* impaired renal function (Creatinine >1.2 mg/dL)
* pregnancy or breast feeding
* inability to obtain informed consent
* active GI Bleeding
* known allergy to Methylene blue or Fluorescein
* participation in other clinical trials within the last 4 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * N=50 patients with unexplained bloating and diarrhoea with suspicion of food intolerance and negative testing with routine methods
  * N=10 patients with Lactose intolerance
  * N=10 patients with Fructose intolerance
  * N=10 volunteers with Barrett's esophagus who need evaluation for possible dysplasia in the Barrett's mucosa with confocal endomicrosopy but no symptoms of bloating and abdominal pain (n=10) to serve as healthy controls for allergy testing
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of mucosal reaction | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Annette Fritscher-Ravens, Prof. Dr., Principal Investigator — University Schleswig-Holstein
Locations (1):
- University Hospital Schleswig Holstein, Campus Kiel, Unit Experimental Endoscopy, Kiel, Germany

REFERENCES:
- [Derived] Fritscher-Ravens A, Schuppan D, Ellrichmann M, Schoch S, Rocken C, Brasch J, Bethge J, Bottner M, Klose J, Milla PJ. Confocal endomicroscopy shows food-associated changes in the intestinal mucosa of patients with irritable bowel syndrome. Gastroenterology. 2014 Nov;147(5):1012-20.e4. doi: 10.1053/j.gastro.2014.07.046. Epub 2014 Jul 30. PMID 25083606